CLINICAL TRIAL: NCT00951275
Title: A Single Arm, Open-label Study of Early Improvement of Anemia and Fatigue During Treatment With Tocilizumab (TCZ) in Combination With DMARDs, in Adult Patients With Moderate to Severe Active Rheumatoid Arthritis.
Brief Title: A Study of Tocilizumab + DMARDs in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22462; 2009-011105-17
Record Dates: First submitted 2009-07-30; First posted 2009-08-04 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Standard DMARDs (Disease Modifying Anti Rheumatic Drugs)

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 6 months
Drug: Standard DMARDs (Disease Modifying Anti Rheumatic Drugs) — As prescribed

SUMMARY:
This single arm study will assess the effect of tocilizumab + DMARDs (Disease Modifying Anti-Rheumatic Drugs)on improvement of anemia and fatigue in patients with moderate to severe active rheumatoid arthritis. Eligible patients who have had an inadequate response to DMARDs will receive tocilizumab 8mg/kg iv every 4 weeks in combination with standard DMARDs, for 6 months. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* rheumatoid arthritis >=6 months duration;
* DAS28>=3.2;
* inadequate response to prior treatment with a stable dose (>=8 weeks) of DMARD therapy.

Exclusion Criteria:

* rheumatic autoimmune disease other than rheumatoid arthritis;
* history of or current inflammatory joint disease other than rheumatoid arthritis;
* unsuccessful treatment with an anti-TNF agent;
* previous/concurrent treatment with any cell-depleting therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2011-07-22 (Actual); Study Completion 2011-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Italy (27):
  - Ospedale Perrino; Medicina Interna - Divisione di Reumatologia, Brindisi, Apulia
  - Presidio Ospedaliero Valle D'itria; Divisione Di Nefrologia, Martina Franca, Apulia
  - Ospedale Galateo; U.O. Di Reumatologia, San Cesario di Lecce, Apulia
  - Azienda Ospedaliera Rummo; Divisione Di Reumatologia, Benevento, Campania
  - Azienda Ospedaliera A. Cardarelli; Medicina III - Divisione di Reumatologia, Napoli, Campania
  - UNIVERSITÀ DI NAPOLI FEDERICO II; Dipartimento di Immunologia Clinica ed Allergologia, Napoli, Campania
  - Ospedale M. Scarlato - Asl Sa1; U.O. Di Reumatologia, Scafati, Campania
  - Irccs Fondazione Salvatore Maugeri-Istituto Scientifico Di Telese;U.O. Riabilitazione Reumatologica, Telese Terme, Campania
  - A.O.U Policlinico S. Orsola Malpighi di Bologna U.O di Medicina Interna Borghi - Pad.2, Bologna, Emilia-Romagna
  - Az. Ospedaliera Univ. di Parma; Medicina Interna e Reumatologia, Parma, Emilia-Romagna
  - Ospedale Guglielmo Da Saliceto Unità Operativa Semplice di Reumatologia e Immunologia, Piacenza, Emilia-Romagna
  - Policlinico Tor Vergata; Divisione Di Reumatologia, Rome, Lazio
  - Ospedale Nuovo Regina Margherita; Divisione di Medicina Interna Reumatologia, Rome, Lazio
  - Ospedale S.Pietro Fatebenefratelli; Divisione di Reumatologia, Rome, Lazio
  - Ospedale Belcolle; Divisione Di Reumatologia, Viterbo, Lazio
  - Ospedale San Paolo; Divisione di Reumatologia, Savona, Liguria
  - ASST PAPA GIOVANNI XXIII; Reumatologia Day Hospital-Torre 2 terzo piano, Bergamo, Lombardy
  - ASST DI MONZA; Reumatologia (Medicina I), Monza, Lombardy
  - IRCCS Istituto Clinico Humanitas; Immunologia Clinica E Reumatologia, Rozzano, Lombardy
  - Ospedale S. Giovanni Bosco; S.C. A Direzione Uni Ria Di Immunologia Clinica, Turin, Piedmont
  - Ospedale Vittorio Emanuele Ii; U.O. Reumatologia Clinica Medica Condorelli, Catania, Sicily
  - A.U.O. G. Martino- Policlinico Univ. Gazzi; Dept. Di Medicina Interna, Divisione Di Reumatologia, Gazzi, Sicily
  - Arnas Ospedale Civico; Medicina Interna II, Palermo, Sicily
  - Az. Osp. Villa Sofia; Unità Operativa Reumatologia, Palermo, Sicily
  - Ospedali Riuniti Villa Sofia- Cervello X; Divisione Medicina I, Palermo, Sicily
  - Ospedale Di Massa; Divisione Di Reumatologia, Massa, Tuscany
  - Ospedale SS Giovanni e Paolo; Divisione Di Reumatologia, Venezia, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) (maximum dose 800 mg) intravenously (IV) once every 4 weeks for a total of 6 infusions.
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg
Started | 105
Completed | 92
Not Completed | 13
Not completed — Administrative Reason | 1
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all enrolled participants who recieved at least 1 dose of study medication.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (maximum dose 800 mg) IV once every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 16

OUTCOME MEASURES:

1. Secondary Outcome: Mean Hemoglobin Levels During the Study
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
g/dL
  Baseline (n=105) | 12.41 (1.51)
  Week 2 (n=99) | 12.84 (1.47)
  Week 4 (n=101) | 12.79 (1.44)
  Week 8 (n=100) | 12.95 (1.45)
  Week 12 (n=94) | 13.06 (1.49)
  Week 16 (n=95) | 13.10 (1.42)
  Week 20 (n=90) | 13.13 (1.40)
  Week 24/End of Study (n=100) | 13.12 (1.39)

2. Primary Outcome: Improvement of Anemia at Week 4 Assessed as Change From Baseline in Hemoglobin
Description: Hemoglobin levels were measured as grams/deciliter (g/dL).
Time Frame: Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 101
g/dL | 0.40 (0.78)

3. Secondary Outcome: Improvement of Anemia Assessed as Change From Baseline in Hemoglobin
Description: Improvement of anemia was evaluated as change in hemoglobin levels from baseline.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
g/dL
  Week 2 (n=99) | 0.47 (0.69)
  Week 4 (n=101) | 0.40 (0.78)
  Week 8 (n=100) | 0.56 (0.95)
  Week 12 (n=94) | 0.64 (1.04)
  Week 16 (n=95) | 0.62 (1.08)
  Week 20 (n=90) | 0.67 (1.10)
  Week 24/End of Study (n=100) | 0.64 (1.20)

4. Secondary Outcome: FACIT-F Scores
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a ≥5-point change from Baseline.
Time Frame: Baseline, Weeks 2, 4, 8,12, 16, 20 and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
units on a scale
  Baseline (n=105) | 28.60 (9.77)
  Week 2 (n=102) | 35.54 (8.53)
  Week 4 (n=101) | 37.24 (8.46)
  Week 8 (n=102) | 39.16 (7.35)
  Week 12 n=94 | 39.02 (8.01)
  Week 16 (n=97) | 40.21 (7.87)
  Week 20 (n=91) | 40.05 (7.77)
  Week 24/End of Study (n=102) | 39.69 (8.39)

5. Secondary Outcome: Improvement of Fatigue Assessed as Change From Baseline in FACIT-F Scores
Description: as for outcome 4
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 102
units on a scale
  Week 2 (n=102) | 7.11 (8.40)
  Week 4 (n=101) | 8.76 (8.83)
  Week 8 (n=102) | 10.74 (9.49)
  Week 12 (n=94) | 10.60 (10.13)
  Week 16 (n=97) | 11.47 (10.24)
  Week 20 (n=91) | 11.63 (10.22)
  Week 24/End of Study (n=102) | 10.84 (11.00)

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Percent (%), 50% or 70% Improvement
Description: The ACR response rates ACR20, ACR50, and ACR70 were defined as ≥20%, ≥50% and ≥ 70% improvement, respectively, in: swollen joint count (SJC) (66 joints) and tender joint count (TJC) (68 joints) and 3 of the 5 remaining ACR parameters: Patient assessment of pain; Patient Global Assessment of Disease Activity; Investigator Global Assessment of Disease Activity; participant self-rated assessment of disability measured by the Health Assessment Questionnaire Disability Index (HAQ-DI); and acute phase response (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]).
Time Frame: Week 24
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
percentage of participants
  ACR20 | 81.0 [73.44 to 88.46]
  ACR50 | 59.0 [49.64 to 68.45]
  ACR70 | 42.9 [33.39 to 52.32]

7. Primary Outcome: Improvement in Fatigue at Week 4 Assessed as Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scores
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a greater than or equal to (≥)5-point change from Baseline.
Time Frame: Week 4
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 101
units on a scale | 8.76 (8.83)

8. Secondary Outcome: Percent Change From Baseline to Week 24 in TJC
Description: Sixty-eight (68) joints were assessed at each visit for tenderness; joints were assessed and classified as tender/not tender. Tender joint count 68 (TJC-68) was calculated as the number of tender joints from 68 joints; the number of tender joints was summed (maximum score 68). Calculated values were used for the analysis. A negative score indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in tender joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 102
percent change in tender joints | -70.65 (47.71)

9. Secondary Outcome: Percent Change From Baseline to Week 24 in SJC
Description: Sixty-six (66) joints were assessed at each visit for swelling; joints were assessed and classified as swollen/not swollen. Swollen joint count 66 (SJC-66) was calculated as the number of swollen joints from 66 joints; the number of swollen joints was summed (maximum score 66). Calculated values were used for the analysis. A negative score indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in swollen joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 100
percent change in swollen joints | -77.59 (31.22)

10. Secondary Outcome: Percent Change From Baseline to Week 24 in Patient Global Assessment of Pain
Description: The participant's assessment of their current level of pain was displayed on a 100-millimeter (mm) horizontal visual analog scale (VAS). The left-hand extreme of the line was described as "no pain" and the right-hand as "unbearable pain". The participant was asked to mark the line that corresponded to their current level of pain; the distance from the left edge was recorded.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 100
percent change in mm | -52.25 (56.88)

11. Secondary Outcome: Percent Change From Baseline to Week 24 in Patient's Global Assessment of Disease Activity
Description: The participant's overall assessment of their current disease activity was displayed on a 100-mm horizontal VAS. The left-hand extreme of the line was described as "no disease activity" (symptom free and no arthritis symptoms) and the right-hand extreme as "maximum disease activity" (maximum arthritis disease activity). Participants were asked to assess their current level of disease activity and mark the line; the distance from the left edge was recorded.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 103
percent change in mm | -55.43 (56.12)

12. Secondary Outcome: Percent Change From Baseline to Week 24 in Investigator's Global Assessment of Disease Activity
Description: The physician's assessment of the participant's current disease activity was displayed on a 100-mm horizontal VAS. The left-hand extreme of the line was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme was considered "maximum disease activity". The physician's global assessment of disease activity was completed by the Efficacy Assessor who could or could not be a physician. The assessor was asked to mark the line corresponding to their assessment of the participant's present level of disease activity; the distance from the left edge was recorded.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 103
percent change in mm | -65.89 (36.72)

13. Secondary Outcome: Percent Change From Baseline to Week 24 in HAQ-DI
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Overall score was computed as the sum of the domain scores and divided by the number of domains answered. Total possible score range was 0-3 where 0 (equals)=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 101
percent change from baseline | -45.94 (54.17)

14. Secondary Outcome: Percent Change From Baseline to Week 24 in High-Sensitivity CRP (Hs-CRP)
Description: hs-CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). hsCRP is measured in milligrams per liter (mg/L).
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in mg/L
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 98
percent change in mg/L | -53.33 (149.9)

15. Secondary Outcome: Percent Change From Baseline to Week 24 in ESR
Description: ESR is a blood test used to monitor therapy in inflammatory diseases such as RA and reflects acute phase reactant levels. ESR is measured in mm per hour (mm/hr); active disease in RA is defined by an ESR greater than 30 mm/hr.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change in mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 98
percent change in mm/hr | -66.00 (47.73)

16. Secondary Outcome: Percentage of Participants With a Response at Week 24 by European League Against Rheumatism (EULAR) Category
Description: Disease response was assessed using EULAR Disease Activity Score Based on 28-Joint Count (DAS28) categories of Good, Moderate, or No Response. Good response was defined as a DAS28 score of less than (<)3.2 and improvement from baseline of >1.2; Moderate response was defined as a DAS28 score of 3.2-5.1 and improvement from baseline of 1.2-0.6 or a DAS28 score of >5.1 and improvement from baseline of >1.2; No response was defined as a DAS28 score of >5.1 and improvement from baseline of <1.2. Participants who discontinued prematurely were identified as non-responders.
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
percentage of participants
  No Response | 12.4 [6.08 to 18.68]
  Moderate Response | 23.8 [15.66 to 31.96]
  Good Response | 63.8 [54.62 to 73.00]

17. Secondary Outcome: Percentage of Participants With a Response at Week 24 by DAS28 Category
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the ESR (mm/hr) and patient's global assessment of disease activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2=low disease activity, DAS28 >5.1=high disease activity and DAS <2.6=remission.
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
percentage of participants
  DAS28 <2.6 | 49.5 [39.96 to 59.09]
  DAS28 ≥2.6 | 50.5 [40.91 to 60.04]

18. Secondary Outcome: Percent Change From Baseline to Week 24 in DAS28 Score
Description: as for outcome 17
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 97
percent change from baseline | -55.78 (23.49)

19. Secondary Outcome: Percentage of Participants With an Improvement of ≥1 g/dL in Hemoglobin
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 105
percentage of participants | 31.4 [22.55 to 40.31]

20. Secondary Outcome: Number of Days as Assessed by Short Form-Health and Labour Questionnaire (SF-HLQ)
Description: The SF-HLQ assessed productivity losses related to health problems in individuals with paid or unpaid work and consists of three modules (absenteeism from paid work, production losses without absenteeism from paid work and hindrance in the performance of paid and unpaid work). Any missed working days or number of worked days with reduced efficiency during the last month were reported.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 25
days
  Missed working days (n=25) | 3.6 (5.0)
  Days with reduced capacity (n=19) | 11.8 (8.8)

21. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Number of Days as Assessed by SF-HLQ
Description: as for outcome 20
Time Frame: Weeks 12 and 24
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 25
days
  Missed working days, Week 12 (n=25) | -3.5 (5.1)
  Days with reduced capacity, Week 12 (n=19) | -4.2 (10.9)
  Missed working days, Week 24 (n=25) | -3.3 (5.1)
  Days with reduced capacity, Week 24 (n=19) | -6.1 (10.7)

22. Secondary Outcome: Number of Hours as Assessed by SF-HLQ
Description: Number of working hours lost, and number of hours of support in in taking over and performing usual household tasks in the last month: chores done by family members, chores done by other persons receiving no pay, home care, other paid care, total number of unpaid hours, and total number of hours during the last month were reported.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 77
hours
  Work lost (n=17) | 13.6 (19.8)
  Chores by family (n=77) | 10.3 (26.5)
  Chores by other unpaid person (n=77) | 0.2 (0.8)
  Home care (n=77) | 0.0 (0.0)
  Other paid care (n=77) | 1.1 (4.2)
  Total unpaid (n=77) | 10.4 (26.5)
  Total (n=77) | 11.5 (26.4)

23. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Number of Hours as Assessed by SF-HLQ
Description: Number of working hours lost, and number of hours of support in in taking over and performing usual household tasks in the last month: chores done by family members, chores done by other persons receiving no pay, home care, other paid care, total number of unpaid hours, and total number of hours during the last month were reported. Changes from baseline were only calculated in participants who completed the questionnaire at all times (baseline, Week 12, and Week 24). Negative number indicates improvement.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 77
hours
  Work lost, Week 12 (n=17) | -8.9 (15.2)
  Work lost, Week 24 (n=17) | -12.1 (20.3)
  Chores by family, Week 12 (n=77) | -4.4 (27.4)
  Chores by family, Week 24 (n=77) | -3.2 (32.0)
  Chores by other unpaid person, Week 12 (n=77) | -0.1 (0.8)
  Chores by other unpaid person, Week 24 (n=77) | -0.2 (0.8)
  Other paid care, Week 12 (n=77) | 1.8 (15.5)
  Other paid care, Week 24 (n=77) | -0.1 (5.1)
  Total unpaid, Week 12 (n=77) | -4.5 (27.3)
  Total unpaid, Week 24 (n=77) | -3.6 (32.0)
  Total, Week 12 (n=77) | -2.7 (31.7)
  Total, Week 24 (n=77) | -3.7 (32.4)

24. Secondary Outcome: SF-HLQ Hindrance Score
Description: Participants were asked if their health problems hindered their paid work on a scale of 1 to 3 (1=no, 2=yes, slightly, 3=yes, very much) and their unpaid work including household work, going shopping, odd jobs, specific activities sharing the household on a scale of 0 to 3 (0=performed without being bothered by healthy problems; 1=performed although bothered by health problems; 2=not performed because of health problems; 3=not performed for reasons other than health problems). The total hindrance score for unpaid work was derived by adding up the item scores. This hindrance score is a measure of the hindrance experienced as a result of health problems during the performance of unpaid work. The minimum score per item for hindrance score was 0, maximum score was 2 (Score of 3 was not considered since the reasons were "other than health problems"). Total score was calculated by adding all 4 items together and ranged from 0 (best possible score) to 8 (worst possible score).
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 85
units on a scale
  Paid work (n=23) | 0.9 (0.5)
  Household work (n=84) | 1.1 (0.5)
  Going shopping (n=84) | 1.0 (0.6)
  Odd jobs (n=84) | 1.1 (0.7)
  Activities for/with children (n=85) | 0.6 (0.6)
  Total score (n=84) | 3.7 (1.7)

25. Secondary Outcome: Change From Baseline to Weeks 12 and 24 SF-HLQ Hindrance Score
Description: Participants were asked if health problems hindered their paid work on a scale of 1 to 3 (1=no, 2=yes, slightly, 3=yes, very much) and their unpaid work including household work, going shopping, odd jobs, specific activities sharing the household on a scale of 0 to 3 (0=performed without being bothered by healthy problems; 1=performed although bothered by health problems; 2=not performed because of health problems; 3=not performed for reasons other than health problems). Hindrance score is a measure of the hindrance experienced as a result of health problems during the performance of unpaid work. The minimum score per item for hindrance score was 0, maximum score was 2 (Score of 3 was not considered since the reasons were "other than health problems"). Total score was calculated by adding all 4 items together and ranged from 0 (best possible score) to 8 (worst possible score). A negative change from baseline indicates improvement.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 85
units on a scale
  Paid work, Week 12 (n=23) | -0.30 (0.70)
  Paid work, Week 24 (n=23) | -0.39 (0.58)
  Household work, Week 12 (n=84) | -0.40 (0.70)
  Household work, Week 24 (n=84) | -0.40 (0.68)
  Going shopping, Week 12 (n=84) | -0.40 (0.64)
  Going shopping, Week 24 (n=84) | -0.40 (0.62)
  Odd jobs, Week 12 (n=84) | -0.38 (0.79)
  Odd jobs, Week 24 (n=84) | -0.36 (0.83)
  Activities for/with children, Week 12 (n=85) | -0.16 (0.69)
  Activities for/with children, Week 24 (n=85) | -0.24 (0.70)
  Total score, Week 12 (n=84) | -1.33 (2.19)
  Total score, Week 24 (n=84) | -1.38 (2.18)

26. Secondary Outcome: Efficiency as Assessed by SF-HLQ
Description: Participants were ask to rate their efficiency in working on a scale of of 0 to 10 (0=very worse, 10=as usual). Overall efficiency score was based on the first 6 items of Question 6, which is a descriptive instrument comprised of 7 items designed to evaluate the specific problems affecting production. These 7 items relate to the effect of health problems on concentration, work pace, the need to be alone, making decisions, postponing and transferring work to others. The participant can choose from 4 possible answers: (almost) never, sometimes, often and (nearly) always. Efficiency score range=6 to 24; higher scores indicate higher impairment.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24
units on a scale
  Efficiency in working (n=21) | 6.3 (2.4)
  Efficiency score (n=24) | 10.1 (3.2)

27. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Efficiency as Assessed by SF-HLQ
Description: Participants were ask to rate their efficiency in working on a scale of of 0 to 10 (0=very worse, 10=as usual). Overall efficiency score was based on the first 6 items of Question 6, which is a descriptive instrument comprised of 7 items designed to evaluate the specific problems affecting production. These 7 items relate to the effect of health problems on concentration, work pace, the need to be alone, making decisions, postponing and transferring work to others. The participant can choose from 4 possible answers: (almost) never, sometimes, often and (nearly) always. Efficiency score range=6 to 24; higher scores indicate higher impairment. Change from baseline was only calculated for participants who completed the questionnaire at all times (baseline, Week 12 and Week 24). A negative change from baseline indicates improvement.
Time Frame: Baseline
Population: ITT population; n=number of participants assessed for the specified parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24
units on a scale
  Efficiency in working, Week 12 (n=21) | 2.0 (2.3)
  Efficiency in working, Week 24 (n=21) | 2.2 (2.4)
  Efficiency score, Week 12 (n=24) | -2.3 (3.0)
  Efficiency score, Week 24 (n=24) | -2.7 (3.0)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected through the entire study period.
Description: Nonserious AEs presented in this record include all AEs reported during the study, not just nonserious events.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/105
Other Adverse Events (participants affected / at risk) | 64/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=105)
Chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=105)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Frequent bowel movements (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Discomfort (General disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Candidiasis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Lipids increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases abnormal (Investigations) | 1
Transaminases increased (Investigations) | 5
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic haemangioma rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Bunion operation (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.